CLINICAL TRIAL: NCT04340609
Title: Allogeneic Umbilical Cord Mesenchymal Stem Cell Therapy for Acute Myocardial Infarction
Brief Title: Stem Cell in Acute Myocardial Infarction
Acronym: AMI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PT. Prodia Stem Cell Indonesia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT/AMI/01/2019
Record Dates: First submitted 2020-02-08; First posted 2020-04-09 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Acute Myocardial Infarction
Keywords: Allogeneic Mesenchymal Stem Cells; Umbilical Cord Mesenchymal Stem Cells; Intravenous Mesenchymal Stem Cells; Intracoronary Mesenechymal Stem Cells

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intravenous Group (Experimental): Dosage of intravenous route is 2 million MSCs/kg for each subject.
  Interventions: Biological: Mesenchymal Stem Cells
- Intracoronary Group (Experimental): Dosage of intracoronary route is ±50 million MSCs for each subject.
  Interventions: Biological: Mesenchymal Stem Cells
- Control Group (No Intervention): Standard treatment of acute myocardia infarction

INTERVENTIONS:
Biological: Mesenchymal Stem Cells — The UC-MSCs from a donor will be cultured in a clinical grade laboratory with xeno-free medium. Maximum passage of expanded-UC MSCs was VI and doubling population is less than 30. To assure the quality of our expanded-UC MSCs at ProSTEM the following tests are done: cell adherence, cell surface marker, in vitro differentiation, cell viability, sterility, Mycoplasma, endotoxin, and karyotyping.
  Arms: Intracoronary Group; Intravenous Group

SUMMARY:
The study will perform UC-MSCs transplantation in 2 groups and 1 control group with standard treatment. Each group consists of 5 subjects. In the first group UC-MSCs will be transplanted via intravenous (IV) route and the second group via intracoronary (IC) route. The IV group will receive 2 million cells/kg for each subject and the dosage of IC group is 50 million cells for each subject. All groups will be observed until 1 year.

ELIGIBILITY:
Inclusion Criteria:

* STEMI patients within 5 days after symptom onset of a first ST-segment elevation myocardial infarction
* Have undergone successful percutaneous coronary intervention (PCI) with drug eluting stent implantation of the infarct-related artery and demonstrated hypokinesia or akinesia that involved more than two thirds of the LV anteroseptal, lateral, or inferior wall with LV ejection fraction of < 45% by echocardiography.
* Ability to understand and provide signed informed consent, or have a designated legal guardian or spouse legally able and willing to make such decisions on the subject's behalf,
* Willingness to attend all scheduled safety follow-up visits
* Subjects need to have a specific criteria of having a single vessel disease (ostial or proximal LAD vessels) that caused extensive anterior infarction (EF <45).

Exclusion Criteria:

* Hemodynamic instability as demonstrated by any of the following,
* Requirement of intra-aortic balloon pump of left ventricular assist device,
* Need for inotropic support (e.g. dopamine and/or dobutamine) for more than 36 hours for the maintenance of mean arterial blood pressure ≥ 60 mmHg,
* Previous or current concomitant serious illnesses, such as cancer, hematological disorders (Hb < 10 g/dL, WBC < 4 or > 11x109/L, or platelets < 100x109/L), kidney failure (creatinine level > 2.5 mg/dL, or creatinine clearance < 30 cc/min), serious infection or any other co-morbidities that could impact patient's short-term survival, psychiatric illness, history of drug of alcohol abuse,
* Prosthetic valves,
* Hypertrophic or restrictive cardiomyopathy,
* Women of child-bearing potential,
* Inability to comply with the protocol,
* Currently using implantable electronic defibrillator or pacemaker

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac events (MACE) endpoints of mortality | 2 weeks after stem cell
  To assess the safety of using allogeneic UC-MSCs therapy for acute myocardial infarction.
Major adverse cardiac events (MACE) endpoints of mortality | 3 months after stem cell
  To assess the safety of using allogeneic UC-MSCs therapy for acute myocardial infarction.
Major adverse cardiac events (MACE) endpoints of mortality | 6 months after stem cell
  To assess the safety of using allogeneic UC-MSCs therapy for acute myocardial infarction.
Major adverse cardiac events (MACE) endpoints of mortality | 12 months after stem cell
  To assess the safety of using allogeneic UC-MSCs therapy for acute myocardial infarction.
Re-infarction | 2 weeks after stem cell
  To assess the safety of using allogeneic UC-MSCs therapy for acute myocardial infarction.
Re-infarction | 3 months after stem cell
  To assess the safety of using allogeneic UC-MSCs therapy for acute myocardial infarction.
Re-infarction | 6 months after stem cell
  To assess the safety of using allogeneic UC-MSCs therapy for acute myocardial infarction.
Re-infarction | 12 months after stem cell
  To assess the safety of using allogeneic UC-MSCs therapy for acute myocardial infarction.
Target vessel revascularization (TVR) | 2 weeks after stem cell
  To assess the safety of using allogeneic UC-MSCs therapy for acute myocardial infarction.
Target vessel revascularization (TVR) | 3 months after stem cell
  To assess the safety of using allogeneic UC-MSCs therapy for acute myocardial infarction.
Target vessel revascularization (TVR) | 6 months after stem cell
  To assess the safety of using allogeneic UC-MSCs therapy for acute myocardial infarction.
Target vessel revascularization (TVR) | 12 months after stem cell
  To assess the safety of using allogeneic UC-MSCs therapy for acute myocardial infarction.
Heart failure hospitalization | 2 weeks after stem cell
  To assess the safety of using allogeneic UC-MSCs therapy for acute myocardial infarction.
Heart failure hospitalization | 3 months after stem cell
  To assess the safety of using allogeneic UC-MSCs therapy for acute myocardial infarction.
Heart failure hospitalization | 6 months after stem cell
  To assess the safety of using allogeneic UC-MSCs therapy for acute myocardial infarction.
Heart failure hospitalization | 12 months after stem cell
  To assess the safety of using allogeneic UC-MSCs therapy for acute myocardial infarction.

SECONDARY OUTCOMES:
Cardiac MRI | 6 months after stem cell
  a test to see improvement in LVEF(%), improvement in regional function, improvement in perfusion, reduction of infarct size.
Cardiac MRI | 12 months after stem cell
  a test to see improvement in LVEF (%), improvement in regional function, improvement in perfusion, reduction of infarct size.
Echocardiography | 6 months after stem cell
  Left ventricular volumes will be determined at end-diastole and end-systole by quantitative biplane assessment. Endocardial borders will be manually traced from apical four-chamber and two-chamber views. Left ventricular volumes will be used to calculate ejection fraction using the biplane modified Simpson's summation-of-disks method recommended by the American Society of Echocardiography.
Echocardiography | 12 months after stem cell
  Left ventricular volumes will be determined at end-diastole and end-systole by quantitative biplane assessment. Endocardial borders will be manually traced from apical four-chamber and two-chamber views. Left ventricular volumes will be used to calculate ejection fraction using the biplane modified Simpson's summation-of-disks method recommended by the American Society of Echocardiography.
Electrocardiography (ECG) | 3 months after stem cell
  to detects cardiac (heart) abnormalities by measuring the electrical activity generated by the heart as it contracts
Electrocardiography (ECG) | 6 months after stem cell
  to detects cardiac (heart) abnormalities by measuring the electrical activity generated by the heart as it contracts
Electrocardiography (ECG) | 12 months after stem cell
  to detects cardiac (heart) abnormalities by measuring the electrical activity generated by the heart as it contracts
Wellness Parameter | 6 months after stem cell
  hs-CRP, antioxidant, IL-6, IL-10, PA1, Fibrinogen
Laboratory Assessment | 12 months after stem cell
  Haematology, Serum Chemistry, Cardiac Biomarker

CONTACTS AND LOCATIONS:
Locations (1):
- PT Prodia StemCell Indonesia, Jakarta, Indonesia